CLINICAL TRIAL: NCT01593202
Title: Long Term Efficacy of Dialectical Behaviour Therapy vs Enhanced Usual Care for Adolescents With Self-Harming and Suicidal Behaviours
Brief Title: Long Term Efficacy of DBT-A in Adolescents With Repetitive Self-harming and Suicidal Behaviours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Mehlum, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES4894
Record Dates: First submitted 2012-04-16; First posted 2012-05-08 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Intentional Self Harm
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialectical behavior therapy (Experimental): Dialectical Behavior Therapy, delivered for 19 weeks, consisted of 1 weekly session of individual therapy (60 minutes), 1 weekly session of multifamily skills training (120 minutes), and family therapy sessions and Telephone coaching with individual therapists outside therapy sessions as needed.
  Interventions: Behavioral: Dialectical behavior therapy
- Enhanced usual care (Active Comparator): Enhanced usual care was 19 weeks of standard care (enhanced for the purpose of the study by requiring that EUC therapists agree to provide on average no less than 1 weekly treatment session per patient throughout the trial) delivered by therapists (4 psychiatrists, 16 clinical psychologists, 6 clinical social workers, 2 clinical pedagogues, 1 specialist nurse, and 1 psychology graduate student) not trained in or practicing DBT.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Dialectical behavior therapy — 16 weeks of Dialectical behavior therapy with one weekly session of individual therapy, one weekly session of multifamily skills training group, telephone coaching and ancillary family therapy and/or pharmacological treatment as needed.
  The treatment has been developed by Marsha Linehan (Linehan, 1993a; 1993b)and adapted for adolescents by Alec Miller (Miller, Rathus & Linehan, 2007). Individual DBT therapists have been trained by drs Alec L Miller and Sarah K Reynolds and have a minimum of one year clinical practise as DBT therapists. The therapists are organised in two consultation teams supervised on a bimonthly basis throughout the entire study by drs Miller and Reynolds respectively.
  Arms: Dialectical behavior therapy
Behavioral: Enhanced usual care — 16 weeks of outpatient treatment in child and adolescent psychiatric clinics in Oslo, on average one weekly session of individual therapy and ancillary supportive. family and/or pharmacological treatment as needed.
  Arms: Enhanced usual care

SUMMARY:
The purpose of the study is to evaluate the long-term efficacy of dialectical behavior therapy (DBT) in treatment of adolescents with deliberate self harm compared to enhanced usual care (EUC). This study follows-up 77 patients in the ages of 12-18 yrs who have been included in an RCT of DBT-A vs EUC. The main inclusion criterion for this study was repetitive self-harm behaviour. The patients were randomly allocated to receive 16 weeks of outpatient DBT or EUC in child and adolescent psychiatric clinics in Oslo. Participants have been assessed so far on five different time-points: baseline (before starting treatment), 9 weeks, 15 weeks, 19 weeks and 71 weeks after start of the treatment. In the current project patients will be assessed a 6th time 2 years after treatment completion.

The main study hypotheses are:

* DBT will be significantly more efficacious in reducing the number of self-harm episodes with or without intent to die, as well as reducing the number of emergency room visits for self-harm or suicidal behaviour, compared to EUC.
* DBT will be significantly more efficacious in reducing the level of suicidal ideation and depressive symptoms compared to EUC.

DETAILED DESCRIPTION:
The study is a long-term follow-up of a randomized trial comparing DBT-A with enhanced usual care (EUC). Participants were randomly allocated to receive either treatment at 1 of the participating child and adolescent psychiatric outpatient clinics in a 1:1 ratio stratified according to gender, presence of major depression, and presence of suicide intent during the most serious episode of self-harm behavior within the 16 weeks before enrollment. Treatment allocation of participants after baseline assessments was based on a permuted block randomization procedure with an undisclosed and variable blocking factor, and daily management of the randomization procedures was performed by an external group. Patients received either DBT or EUC by therapists working at and funded by the 10 child and adolescent psychiatric outpatient clinics participating in the study. They were assessed during treatment (9 and 15 weeks), at treatment completion 19 weeks, and at 71 weeks. In this study they are assessed at 2 years after treatment completion.

The assessment of outcomes include: number of self-reported self-harm episodes (suicide attempts and non-suicidal self-harm episodes combined, measured by Lifetime Parasucide Count); the severity of suicidal ideation as measured by the 15-item self-report Suicidal Ideation Questionnaire (SIQ-JR; and level of depressive symptoms as measured by the 13-item version of the self-report Short Mood and Feelings Questionnaire (SMFQ) and through the interviewer rated 10-item Montgomery-_Asberg Depression Rating Scale (MADRS). Other outcomes are hopelessness, measured by the 20-item self-report Beck Hopelessness Scale (BHS);borderline symptoms, assessed through the 23-itemself-report Borderline Symptom List (BSL); Borderline Personality Disorder as measured by SCID-II; and hospital admissions and emergency department visits because of self-harm.

ELIGIBILITY:
Inclusion Criteria:

Patients included in the initial RCT 'Treatment for Adolescents With Deliberate Self Harm' (ClinicalTrials ID NCT00675129). Inclusion criteria for this study were:

* History of repeated deliberate self harm (last episode within last months)
* Satisfies at least 2 criteria of DSM-IV Borderline Personality Disorder (as measured by SCID-II) in addition to the self-destructive criterion.

Or: Satisfies at least 1 criterion + 2 criteria scored below threshold (score 2) of DSM-IV Borderline Personality Disorder (as measured by SCID-II) in addition to the self-destructive criterion.

Exclusion Criteria:

* Psychotic disorders
* Anorexia Nervosa
* Substance dependence disorder
* Mental retardation (IQ less than 70)
* Asperger syndrome/autism

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2012-01; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of subsequent episodes of deliberate self harm and time elapsed to future episodes of deliberate self harm | 2 years after end of treatment
  Measured by the Linehan Parasuicide Count (LPC)

SECONDARY OUTCOMES:
Severity of suicidal ideation | 2 years
  Measured by the Suicidal Ideation Questionnaire Jr (SIQ-Jr). Scale range: min= 0, max = 90. High values represent a worse outcome.
Frequency of subsequent emergency room visits, hospitalizations and use of additional treatments due to risk of deliberate self-harm behavior | 2 years
  Measured through and interview specifically developed for the purpose and through linkage with the Norwegian Patient Register
Self reported level of depressive symptoms | 2 years
  Measured by the Moods and feelings questionnaire (MFQ). Scale range: min = 0, max = 26. High levels represent a worse outcome
Researcher rated level of depressive symptoms | 2 years
  Measured through the Montgomery Asberg Depression Rating Scale (MADRS). Scale range: min = 0, max = 60. High levels represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Mehlum, Professor, Principal Investigator — National Centre for Suicide Research and Prevention
Locations (1):
- National Centre for Suicide Research and Prevention Unit/University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehlum L, Ramleth RK, Tormoen AJ, Haga E, Diep LM, Stanley BH, Miller AL, Larsson B, Sund AM, Groholt B. Long term effectiveness of dialectical behavior therapy versus enhanced usual care for adolescents with self-harming and suicidal behavior. J Child Psychol Psychiatry. 2019 Oct;60(10):1112-1122. doi: 10.1111/jcpp.13077. Epub 2019 May 25. PMID 31127612
- See also: Information about the research project in Norwegian — http://www.med.uio.no/klinmed/forskning/sentre/nssf/forskning/nssf-prosjekter/dbt-langtidseffekt/